CLINICAL TRIAL: NCT00673972
Title: A Comparative Study of Epigastric Pain Syndrome and Postprandial Distress Syndrome in Personality, Helicobacter Pylori Infection, Gastric Emptying and Response to Lansoprazole Treatment
Brief Title: Comparative Study of Epigastric Pain Syndrome and Postprandial Distress Syndrome
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: difficulty in recruiting patients
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Ming-Shiang Wu, National Taiwan University Hospital
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 200705051M
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2010-03-10 (Estimated); Status verified 2010-03

CONDITIONS: Functional Dyspepsia; Epigastric Pain Syndrome; Post Prandial Distress Syndrome
Keywords: Functional dyspepsia; Gastric emptying; Helicobacter pylori; Lansoprazole; Epigastric pain syndrome; Postprandial distress syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPS (Active Comparator): Patients with functional dyspepsia will be classified into EPS or PDS two subgroups according to Rome III diagnostic criteria.
  Interventions: Radiation: gastric scintigraphy
- PDS (Active Comparator): Patients with functional dyspepsia will be classified into EPS or PDS two subgroups according to Rome III diagnostic criteria.
  Interventions: Radiation: gastric scintigraphy

INTERVENTIONS:
Radiation: gastric scintigraphy — All tests start after overnight fast. Test meals consists of 120g scrambled egg, two slices of toasted bread, 30g of strawberry jam and 120ml of water. 12MBg (0.33mCi) of 99mTc sulfur colloid is mixed with egg thoroughly before the mixture cooked in a microwave oven for 2 minutes. All meals are prepared on the morning of examination and consumed within 20 minutes.
  Anterior and posterior images of the gastric region are taken within one minute after completion of test meals. Subsequent images are taken every 2 minutes in the first 60 minutes and at 120 minutes and 180 minutes. One-min images of gastric region at upright position are taken in the 140keV 99mTc peak with a 20% window.
  Other Names: gastric emptying time

SUMMARY:
The purpose of this study is to compare postprandial distress syndrome and epigastric pain syndrome in demographics psychological features, infection of Helicobacter pylori, gastric emptying and therapeutic response to lansoprazole.

DETAILED DESCRIPTION:
Functional dyspepsia is a common clinical disorder with significant impact on quality of life and with enormous social cost. Previous studies have revealed that functional dyspepsia is not a homogenous disease but a heterogenous symptom complex. Because of heterogeneity in etiology and pathogenesis, no specific treatment is appropriate for all patients with functional dyspepsia. Currently available treatments demonstrated efficacy only in subsets of patients.

Appropriate subgrouping of functional dyspepsia, which categorizes more homogenous patients into the same group, will correlate better with specific etiologic factors and pathogenetic mechanisms. Consequently patients may have appropriate specific treatment based on more directed pathologenesis and subgrouping. To this end, American Gastroenterology Association launched new edition of clinical guide for functional gastrointestinal disorder, the Rome III in May 2006. The new diagnostic criteria of Rome III de-emphasized functional dyspepsia as an entity and recommended sub-classification into two conditions: postprandial distress syndrome and epigastric pain syndrome. However whether this new diagnostic criteria and systems are effective and clinically relevant remains unknown.

Aims:

We aim to compare postprandial distress syndrome and epigastric pain syndrome in demographics psychological features, infection of Helicobacter pylori, gastric emptying and therapeutic response to lansoprazole.

ELIGIBILITY:
Inclusion Criteria:

* aged greater than 20 years
* fulfill Rome III diagnostic criteria

Exclusion Criteria:

* children and teenagers aged less than 20 years
* Organic lesions such as ulcers, tumors, bleeding, vasculopathy or esophagitis as demonstrated on upper endoscopy
* concurrent illness with malignancy, diabetes mellitus, liver cirrhosis, renal failure or porphyria
* diagnosis of organic disease for dyspeptic symptoms by treating physicians
* history of abdominal surgery
* concurrent user of aspirin and NSAID
* history of allergy or severe side effects to lansoparzole
* pregnant or lactating women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-11 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Primary end point of the study is to compare the gastric emptying time in epigastric pain syndrome and that in postprandial distress syndrome | After four-week treatment of lansoprazole

SECONDARY OUTCOMES:
Psychiatric distress, personality traits, infection of H. pylori and symptom improvement to lansoprazole | after four-week treatment of lansoprazole

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, M.D.PHD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan